CLINICAL TRIAL: NCT05171608
Title: Preoperative Ultrasound-based Protocol for Optimization of Fluid Therapy to Prevent Hypotension Associated to General Anesthesia: a Randomized Controlled Trial
Brief Title: Preoperative Ultrasound-based Protocol for Optimization of Fluid Therapy to Prevent Early Intraoperative Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Marcell Szabo, assistant lecturer, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PUSPO
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Anesthesia; Hypotension; Lung Ultrasound; Echocardiography; Perioperative Complication
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The attending anesthesiologist, participant and outcomes assessors will be blinded to randomization and result of preoperative ultrasound scans. The attending anesthesiologist (not aware of randomization and ultrasonographic findings) gives a dose recommendation for fluid therapy for all patients. The investigator will be aware of the randomization and ultrasound results. This investigator will choose the fluid therapy (conforming to the ultrasound based protocol OR to the dose-recommendation of the attending anesthesiologist) following the results of randomization and ultrasound scans in the USP group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-based protocol group (USP) (Experimental): Preoperative intravenous (IV) fluid therapy is order according to the result of the preoperative ultrasound scans of the inferior vena cava and the lungs (2 hours and 30 minutes before surgery)
  Interventions: Procedure: Ultrasound-based protocol based fluid therapy
- Conventional fluid therapy (No Intervention): Preoperative IV fluid therapy (isotonic, balanced crystalloid infusion, if any) is determined by the discretion of the attending anesthesiologist.

INTERVENTIONS:
Procedure: Ultrasound-based protocol based fluid therapy — Protocol of the interventional group according to the ultrasonographic findings:
  Ultrasound scan 2 hours before surgery:
  IVCCI>40 percent and absence of symmetric anterior 'B-profile' on the lung ultrasound indicate intravenous (IV) fluid therapy: 8 ml/kg of isotonic, balanced crystalloid infusion.
  IVCCI≤40 percent AND/OR symmetric anterior 'B-profile' contraindicates further IV fluid therapy.
  A 2nd ultrasound scan at 30 minutes before surgery:
  IVCCI>40 percent and absence of symmetric anterior 'B-profile' on the lung ultrasound indicate further IV fluid therapy: 5 ml/kg of isotonic, balanced crystalloid infusion.
  IVCCI≤40 percent AND/OR symmetric anterior 'B-profile' contraindicates further IV fluid therapy.
  Arms: Ultrasound-based protocol group (USP)

SUMMARY:
Background: Intraoperative hypotension increases 30-day mortality and the risks of myocardial injury and acute renal failure. Patients with inadequate volume reserve before the induction of anesthesia are highly exposed. The identification of latent hypovolemia is therefore crucial. Ultrasonographic measurement of the inferior vena cava collapsibility index (IVCCI) is able to detect volume responsiveness in circulatory shock and growing evidence support the theory that higher IVCCI can predict intraoperative hypotension.

The aim of the present study is to evaluate the potential benefit of an ultrasound-based protocol for preoperative fluid optimization. The investigators will perform a randomized-controlled study involving elective surgical patients. An ultrasound-based protocol (USP) arm and a conventional fluid therapy group (CFT) are to be formed. Ultrasound examinations will be performed twice in both groups: 2 hours and 30 minutes preoperatively. The inferior vena cava and the anterior lung fields will be scanned. In the USP group the participants will receive fluid therapy according to the ultrasonographic findings: high level of IVCCI and absence of signs of pulmonary edema will indicate fluid therapy. In the CFT group the attending anesthesiologist (blinded to the results of ultrasonography) will order fluid therapy on the basis of daily routine and clinical judgement.

The investigators will evaluate the incidence of intraoperative hypotension (primary outcome), postoperative metabolic status and organ functions and the amount of the administered intravenous fluids in both groups.

DETAILED DESCRIPTION:
A randomized-controlled study with 80 participants.

The investigators will use computer-generated unpaired random allocation method to an ultrasound-based protocol (USP) group or to the conventional fluid therapy (CFT) group.

Preoperative ultrasound examinations will be performed twice in both groups: 2 hours and 30 minutes preoperatively. The inferior vena cava and the lung fields (so called BLUE - Bedside Lung Ultrasound in Emergency - points: 2nd or 3rd intercostal space anterior, 5th-6th interspace anterior and posterior axillary line position) will be scanned. The collapsibility index (IVCCI) of the IVC is calculated, >40 percent is considered 'high IVCCI'. Lung ultrasound (LUS) is evaluated as indicative for 'lung congestion' if symmetric anterior B-profiles (at least 3 B-lines in anterior lung fields) are detected.

Baseline demographic (age, sex, height, weight) and comorbidity data (history of hypertension, chronic heart failure, coronary or cerebrovascular disease, respiratory illness e.g. COPD, past COVID, diabetes on insulin treatment) together with laboratory data (haemoglobin, creatinine, blood urea) are to be recorded.

A standardized practice of monitoring and induction of general anesthesia will allow for the detection of immediate and early (first 10 minutes of anesthesia) hypotensive events. A follow up for 24 hours is necessary for evaluating the fulfillment of secondary endpoints. A semi-quantitative lung ultrasound after 24 hours will estimate lung aeration.

ELIGIBILITY:
Inclusion Criteria:

Elective surgery

* General surgical procedures
* Estimated duration of anesthesia > 60 minutes
* ASA class 2 or 3

Exclusion Criteria:

* Emergency procedure
* Reoperation, redo procedure
* Patient who is incapable of acting
* Uncontrolled hypotension (<90 mmHg)
* Uncontrolled hypertension (>180 mmHg)
* High risk valvular disease (Aortic Stenosis)
* Endocrine hypertension (Conn's syndrome, phaeochromocytoma)
* Sepsis (infection and SOFA≥2 pt)
* Conditions blocking lung ultrasound (pneumothorax without drainage, former pulmonary resection, pleural effusion affecting more than 2 interspaces)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of hypotension associated to general anesthesia induction | first 10 minutes of anesthesia
  mean arterial pressure < 65 mmHg AND/OR ≥30 percent of decrease compared to baseline (before induction of anesthesia)

SECONDARY OUTCOMES:
Dose of preoperative fluid therapy (in millilitres) | preoperative time frame on the day of surgery
  intravenous fluid therapy before anesthesia induction
Dose fluid therapy of the operative day (in millilitres) | 24 hours
  all intravenous fluid therapy on the day of surgery
lactate level (mmol/l) | 1st postoperative hour
  highest lactate level in mmol of an arterial blood sample
base excess (mmol/l) | 1st postoperative hour
  worst base excess level in mmol of an arterial blood sample
urine output (millilitres/24 h) | 24 hours
  summarized urine output after surgery
lung ultrasound score (LUS) | 24th postoperative hour
  Summarized lung ultrasound score of 12 fields of the thorax (0-36 pts)

CONTACTS AND LOCATIONS:
Overall Officials: Sándor Soós, PhD, Principal Investigator — Semmelweis University, Department of Surgery, Transplantation and Gastroenterology
Locations (1):
- Semmelweis University, Deparment of Surgery, Transplantation and Gastroenterology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szabo M, Bozo A, Darvas K, Horvath A, Ivanyi ZD. Role of inferior vena cava collapsibility index in the prediction of hypotension associated with general anesthesia: an observational study. BMC Anesthesiol. 2019 Aug 7;19(1):139. doi: 10.1186/s12871-019-0809-4. PMID 31390983
- [Background] Szabo M, Bozo A, Darvas K, Soos S, Ozse M, Ivanyi ZD. The role of ultrasonographic lung aeration score in the prediction of postoperative pulmonary complications: an observational study. BMC Anesthesiol. 2021 Jan 14;21(1):19. doi: 10.1186/s12871-021-01236-6. PMID 33446103
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Lichtenstein DA. BLUE-protocol and FALLS-protocol: two applications of lung ultrasound in the critically ill. Chest. 2015 Jun;147(6):1659-1670. doi: 10.1378/chest.14-1313. PMID 26033127
- [Background] Zhang J, Critchley LA. Inferior Vena Cava Ultrasonography before General Anesthesia Can Predict Hypotension after Induction. Anesthesiology. 2016 Mar;124(3):580-9. doi: 10.1097/ALN.0000000000001002. PMID 26771910
- [Derived] Szabo M, Pleck AP, Soos SA, Keczer B, Varga B, Szell J. A preoperative ultrasound-based protocol for optimisation of fluid therapy to prevent early intraoperative hypotension: a randomised controlled study. Perioper Med (Lond). 2023 Jun 27;12(1):30. doi: 10.1186/s13741-023-00320-4. PMID 37370150